CLINICAL TRIAL: NCT06586658
Title: An Exploratory Clinical Study of the Safety and Efficacy of Anti-CD70-CAR-T Cell Injection in Patients With Locally Advanced or Relapsed/Metastatic Renal Cell Carcinoma With CD70+ Inoperable
Brief Title: Anti-CD70-CAR-T Cell Injection for the Treatment of Locally Advanced or Relapsed/Metastatic CD70+ Inoperable Renal Cells
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Shanghai First Song Biotechnology Co., LTD (Industry)
Responsible Party: Principal Investigator, Ren Shancheng, Professor, Chief of Urology, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD70-CN-A5
Record Dates: First submitted 2024-08-07; First posted 2024-09-19 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Renal Cell Carcinoma
Keywords: CART; CD70; Renal carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental)
  Interventions: Biological: anti-CD70-CAR-T cells

INTERVENTIONS:
Biological: anti-CD70-CAR-T cells — The subjects received infusions of anti-CD70 CART cells following completion of lymphodepleting preconditioning chemotherapy. Dosage: 3×10^6 cells/Kg; 1×10^7 cells/Kg; 2×10^7 cells/Kg.

SUMMARY:
This is an investigator-initiated trial to evaluate the role of anti-CD70-CAR T cells in locally advanced or recurrent/metastatic renal cell carcinoma that is inoperable.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the role of anti-CD70-CAR T cells in locally advanced or recurrent/metastatic renal cell carcinoma that is inoperable

Study intervention consists of a single infusion of CAR-transduced autologous T cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

Interim analysis will be performed when the last participant finishes the visit of 12 weeks after CAR-T cells infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign informed consent, and voluntarily participate in clinical research;
2. Age ≥18, and <70 years old, gender is not limited;
3. Histopathologically or cytologically confirmed advanced malignant renal cell carcinoma of CD70+ with at least VEGFR-targeted therapy and an immune checkpoint therapy (either combination therapy or sequential therapy);
4. At least one measurable lesion with a maximum diameter of less than 6 cm according to RECIST 1.1;
5. Expected survival ≥12 weeks;
6. ECOG score ≤2 points;
7. Have sufficient hematologic function and have not received blood transfusion or cell growth factor therapy within 7 days prior to the hematologic evaluation during the screening period (2 weeks interval is required for those receiving long-acting agents such as PEG-rhG-CSF, allowing the use of recombinant erythropoietin) :

   * Neutrophil absolute value ≥1.5×109/L
   * Hemoglobin ≥80g/L
   * Platelets ≥75×109/L
   * Lymphocytes (ALC) ≥0.3×109/L
8. Adequate liver function: serum total bilirubin ≤1.5× upper limit of normal (ULN) (for Gilbert syndrome patients, total bilirubin ≤3×ULN), aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN; If there is liver metastasis, allow AST, ALT≤5×ULN);
9. Adequate renal function: creatinine ≤1.5×ULN or endogenous creatinine clearance ≥50 mL/min (using Cockcroft Gault formula);
10. Left ventricular ejection fraction (LVEF) of echocardiography was ≥50%.
11. There was no evidence of dyspnea at rest and pulse oximetry was >93% without oxygen.
12. Activated partial thromboplastin time (APTT) ≤1.5×ULN and International normalized ratio (INR) ≤1.5×ULN;
13. Good venous access (for apheresis) and no other contraindications for blood cell separation;
14. Pregnancy tests for women of childbearing age must be negative. All subjects must agree to use an effective contraceptive method at the same time from the time of signing the informed consent to 12 months after the final administration of the study drug.

Exclusion Criteria:

Patients are not eligible to participate in this trial if they meet any of the following conditions:

1. Previous use of any CAR T cell products or other genetically modified T cell therapy;
2. Patients who have a history of allogeneic stem cells or solid organ transplantation or are waiting for organ transplantation;
3. Patients with acute or uncontrolled active infection who currently require intravenous anti-infective therapy, and patients taking antibiotics to prevent infection should be allowed to participate in the study at the discretion of the investigator;
4. Active hepatitis B (hepatitis B surface antigen positive and hepatitis B DNA>103 copies /mL or >200IU/mL), active hepatitis C (hepatitis C antibody positive and RNA positive); Active syphilis infection (RPR or TRUst-positive), human immunodeficiency virus (HIV) infection (HIV positive);
5. Patients with low sodium and/or hypokalemia with blood sodium <125mmol/L and/or blood potassium <3.5mmol/L (unless sodium and/or potassium supplementation is required prior to study participation to restore blood sodium and/or potassium above this level);
6. Imaging results showed that the proportion of liver replaced by tumor was ≥50%;
7. There was clinically uncontrollable third space effusion, which was judged by the researcher not suitable for inclusion;
8. Previously received anti-CD70 therapy;
9. Receiving continuous systemic steroid medication (prednisone > 10mg/ day or equivalent dose of other hormones) within 14 days of preapheresis or 3 days before cell therapy, except for recent or current topical steroid use;
10. Toxicity from previous antitumor therapy has not recovered (>CTCAE version 5.0 Grade 1), except for alopecia, pigmentation, and other tolerable events as determined by the investigator or laboratory abnormalities permitted under the protocol;
11. The eluting period of preaphermative antitumor therapy met the following requirements:

    * ≦2 weeks or 5 half-lives of chemotherapy, small molecule targeted therapy, radiotherapy, endocrine therapy, immunomodulatory therapy, and Chinese medicine with anti-tumor indications
    * ≦4 weeks of macromolecular targeted therapy and immunotherapy
    * ≦4 weeks of anti-tumor vaccine
    * ≦4 weeks of investigational medication/therapy
12. Previous or current co-occurrence of other malignancies (other than basal cell carcinoma of the skin, carcinoma in situ of the breast/cervix and other malignancies that have been cured or are free of disease and have not been treated in the past five years);
13. Previous history of primary or secondary tumors of the central nervous system (CNS) (except stable ≥4 weeks after treatment, no current CNS related signs and no drug control ≥14 days);
14. Patients with other central nervous system diseases (such as seizures, cerebral hemorrhage, dementia, etc.) that researchers have judged may affect the safety of subjects;
15. Uncontrolled hypertension (systolic blood pressure ≥150 MMHG and/or diastolic blood pressure ≥95mmHg after standard treatment), unstable angina, congestive heart failure of New York Heart Association grade III or higher, or significant abnormalities on ECG, Severe arrhythmias requiring treatment and a history of myocardial infarction within 6 months prior to initiation of study therapy;
16. Patients with severe respiratory diseases, such as interstitial lung disease, active pulmonary tuberculosis, and patients who have received extensive radiation therapy in the lung, were not considered suitable for inclusion by researchers;
17. Patients with active or past autoimmune diseases with the possibility of recurrence (e.g. systemic lupus erythematosus, rheumatoid arthritis, etc.), except for type 1 diabetes, hypothyroidism requiring hormone replacement therapy, skin diseases without systemic treatment (e.g. vitiligo, psoriasis or alopecia);
18. In the investigator's judgment, any serious or uncontrollable systemic disease, systemic comorbiditis, other serious comorbiditis (such as hemophagic cell syndrome, etc.), or special conditions of the tumor may make the patient unfit to enter the study or affect protocol compliance, or significantly interfere with the correct evaluation of the safety, toxicity, and effectiveness of the investigatory drugs;
19. Had any major surgery (other than exploratory laparotomy or laparoscopic exploration) or severe trauma within 4 weeks prior to apheresis, had major surgery scheduled during DLT observation, or had not fully recovered from any previous invasive procedure;
20. Patients who are allergic to or intolerant to antisepsis agents that may be used during the study or to medications that are appropriate for the treatment of CRS, including but not limited to fludarabine and cyclophosphamide or toluzumab; Known to be allergic to anti-CD70-CAR-T ingredients; Or have any history of severe allergies, such as anaphylactic shock;
21. Women who are pregnant, who plan to become pregnant during the trial, or who are breastfeeding;
22. Patients judged by the investigator to be unable or unwilling to comply with clinical protocols;
23. Persons involved in the planning and execution of the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2027-07-16 (Estimated); Study Completion 2027-07-16 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) within 28 days after infusion | Within 28 days after infusion
Incidence and severity of adverse events after infusion (including abnormal test values, physical examination, vital sign parameters) | 1 year
Maximum tolerated dose (MTD) or recommended dose in subsequent clinical trials | Up to 28 days from CAR-T infusion

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of CAR-T infusion until date of first documented progression or date of death from any cause, whichever came first, assessed up to 15 years
  Progression-free survival (PFS) is the time between the date of first administration and the date of tumor progression (PD as assessed by imaging diagnosis) or the date of all-cause death (whichever occurs first).
Overall survival (OS) | From date of CAR-T infusion until date of death from any cause, assessed up to 15 years
  Overall survival (OS) is the time between the date of first dosing and the date of all-cause death.
Duration of efficacy (DOR) | Through study completion, an average of 1 year
  Duration of efficacy (DOR) is the time between meeting the criteria for treatment effectiveness (first recorded complete or partial response) and the first clear recurrence or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Shancheng Ren, MD,PhD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Changzheng hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to concerns regarding the security of patient personal information.